CLINICAL TRIAL: NCT04714177
Title: Efficacy and Safety of Edaravone Dexborneol in Addition to Standard of Care in Patients With Hypertensive Intracerebral Hemorrhage: a Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Edaravone Dexborneol for Treatment of Hypertensive Intracerebral Hemorrhage
Acronym: ED-ICH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jinsheng Zeng, MD, PhD, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIM23-ICH-201
Record Dates: First submitted 2021-01-15; First posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Edaravone Dexborneol (Experimental): Edaravone Dexborneol injection
  Interventions: Drug: Edaravone Dexborneol
- Placebo (Placebo Comparator): Edaravone Dexborneol matching injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Edaravone Dexborneol — Edaravone Dexborneol 37.5 mg, containing Edaravone 30 mg and Dexborneol 7.5 mg, Edaravone Dexborneol 37.5 mg BID, 14 days, addition to standard of care of Intracerebral Hemorrhage
  Arms: Edaravone Dexborneol
Drug: Placebo — Edaravone Dexborneol matching injection, addition to standard of care of Intracerebral Hemorrhage
  Arms: Placebo

SUMMARY:
pending

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent from the patient or legally acceptable representative
* Males and females
* Diagnose as hypertensive intracerebral hemorrhage
* Onset of symptoms within 6~48 hours
* Position of bleeding major in basal ganglia
* The sum of scores on items 5 and 6 on the NIHSS were >= 2 at baseline and the total score (items 1-11) was >=6 and <=20
* Volume of Hematoma <= 30 ml
* Premorbid mRS score of 0 or 1

Exclusion Criteria:

* Allergy to known study drugs or excipients
* Experienced stroke in latest 3 month
* Volume of Hematoma > 5 ml in other bleeding position
* Obstructive hydrocephalus
* Any diagnosis as other than hypertensive ICH
* Unconsciousness
* Severe concurrent illness with life expectancy less than 90 days
* Pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
The proportionof Participants With modified Rankin Scale (mRS) 0 ~ 1 | 90 days after the first dose of study treatment

SECONDARY OUTCOMES:
The proportion of death | 90 days after the first dose of study treatment
The proportionof Participants With modified Rankin Scale (mRS) | 14, 30 and 90 days after the first dose of study treatment
The change in the NIH stroke scale (NIHSS) from the baseline | 14, 30 and 90 days after the first dose of study treatment
The proportionof Participants With Glasgow Outcome Score (GOS) | 14, 30 and 90 days after the first dose of study treatment
Barthel Index (BI) | 90 days after the first dose of study treatment
Stroke Specific Quality of Life Scale (SS-QOL) | 90 days after the first dose of study treatment